CLINICAL TRIAL: NCT03024944
Title: TAU PET Imaging in Northern Manhattan Study of Metabolism and Mind
Acronym: TAUPET
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 18F-THK5351 was reported non-specific binding of MAO receptors.
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, José A. Luchsinger, Associate Professor of Medicine and Epidemiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR1419; 3R01AG050440 (NIH)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus; Alzheimer Dementia
Keywords: Diabetes Mellitus; Alzheimer's Disease; Dementia; THK
MeSH Terms: conditions — Diabetes Mellitus; Alzheimer Disease; Dementia | interventions — THK5351

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brain Imaging with 18F-THK-5351 (Experimental): This group consists of 30 adult subjects: 10 with Type 2 diabetes, 10 with pre-diabetes, and 10 with normal glucose tolerance. Each subject will receive a baseline scan and a follow-up PET scan with 18F-THK-5351.
  Interventions: Drug: 18F-THK-5351

INTERVENTIONS:
Drug: 18F-THK-5351 — Intravenous (IV) catheter (tube) placed in participant arm. A small amount of 18F-THK-5351 will be injected into the IV enough time has passed for this contrast to collect in the tissue in the brain (approximately one half-hour), and participant will lie on a bed which slides into a PET Scanner to complete Tau imaging.
  Other Names: THK

SUMMARY:
The purpose of this project is to study brain imaging of a substance called tau, which is found in brains of persons with Alzheimer's disease, using the Tau binder, 18F-THK-5351, for live imaging of tau in the brain. The main goal of this proposal is to study whether diabetes status (type 2 diabetes [referred to as diabetes] and pre-diabetes, compared with normal glucose tolerance [NGT]), is associated with increased tau accumulation in the brain, one of the culprits of Alzheimer's disease, in a community-based group of middle aged Caribbean-Hispanics with a mean age of 63 years. The investigators propose to conduct tau positron emission tomography (PET) imaging in 30 middle aged Hispanics.

DETAILED DESCRIPTION:
The burden of late onset Alzheimer's dementia (LOAD) and its antecedents is increasing without known prevention or cure, and diabetes seems to be one of the strongest risk factors. The predominating causal model in Alzheimer's disease (AD) research is based on the amyloid hypothesis, which posits that amyloid (A) deposition in the brain causes synaptic dysfunction resulting in early memory deficits and progression to mild cognitive impairment (MCI) and dementia. Tau has also gained increasing interest as an AD pathology feature, biomarker, and treatment target.

There are no known curative or preventive measures for LOAD. One of the strongest potential LOAD risk factors is type 2 diabetes, an abnormal elevation of blood glucose associated with microvascular and macrovascular complications including cerebrovascular disease. Many studies have reported an association of diabetes with dementia, including LOAD and vascular dementia (VD). Most studies have found that diabetes is associated with an increased risk of both LOAD and VD, with a stronger association for VD compared with LOAD. Thus, this study focuses on the relation of diabetes, pre-diabetes, and elevated glucose, with AD.

ELIGIBILITY:
Inclusion Criteria:

* All persons who have undergone magnetic resonance imaging (MRI) and amyloid PET already, or those who prospectively are deemed eligible for the parent study covered under protocol AAAQ2950, will be approached for participation.

Exclusion Criteria:

* Person who are not participating in the MRI and amyloid PET under protocol AAAQ2950

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Amount of Tau Accumulation by Measuring Standardized Uptake Value Ratio (SUVR) | 2 Years
  The primary aim is to measure 18THK-5351 binding (SUVR) in medial temporal and inferior temporal cortex, cross-sectionally and longitudinally.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Luchsinger, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided